CLINICAL TRIAL: NCT01663844
Title: New Clinical Applications for Internet-based Cognitive Behavior Therapy: An Adaptive Treatment Strategy to Decrease the Number of Failed Treatments, and a Combination Treatment for Insomnia and Depression.
Brief Title: New Clinical Applications for Internet-based Cognitive Behavior Therapy for Insomnia and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Viktor Kaldo, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012/934-31/4
Record Dates: First submitted 2012-08-03; First posted 2012-08-13 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Insomnia; Major Depression; Minor Depression
Keywords: Cognitive behavior therapy; Internet treatment; Self-help treatment; Insomnia; Depression; ICBT; CBT-i; CBT-d
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- (Study 1) ICBT for insomnia and depression (Experimental)
  Interventions: Behavioral: Therapist guided Internet-CBT for insomnia and depression
- (Study 1) ICBT for depr. plus placebo insomnia intervention (Active Comparator)
  Interventions: Behavioral: Therapist Guided Internet-CBT for depression plus insomnia placebo
- (Study 2) ICBT for insomnia with added support (Experimental)
  Interventions: Behavioral: Therapist guided Internet-CBT for insomnia w. extra support
- (Study 2) ICBT for insomnia with regular level of support (Active Comparator)
  Interventions: Behavioral: Therapist guided Internet-CBT for insomnia

INTERVENTIONS:
Behavioral: Therapist guided Internet-CBT for insomnia w. extra support — (Study 2) A 9 week long, structured self-help program with weekly reports to, and feedback from, a CBT therapist over the Internet. Includes traditional CBT-methods for insomnia plus extra therapist support.
  Arms: (Study 2) ICBT for insomnia with added support
Behavioral: Therapist guided Internet-CBT for insomnia — (Study 2) A 9 week long, structured self-help program with weekly reports to, and feedback from, a CBT therapist over the Internet. Includes traditional CBT-methods for insomnia. Regular therapist support.
  Arms: (Study 2) ICBT for insomnia with regular level of support
Behavioral: Therapist guided Internet-CBT for insomnia and depression — (Study 1) A 12 week long, structured self-help program with weekly reports to, and feedback from, a CBT therapist over the Internet. Includes traditional CBT-methods for insomnia and depression.
  Arms: (Study 1) ICBT for insomnia and depression
Behavioral: Therapist Guided Internet-CBT for depression plus insomnia placebo — (Study 1) A 12 week long, structured self-help program with weekly reports to, and feedback from, a CBT therapist over the Internet. Includes traditional CBT-methods for depression. A placebo intervention for insomnia is added.
  Arms: (Study 1) ICBT for depr. plus placebo insomnia intervention

SUMMARY:
This study includes two sub-trials. Both are included in this singe registration since they have parallel inclusion of participants and have been approved by the Swedish ethics board together in one application.

Trial 1 includes patients with both insomnia and major or minor depression. Participants are randomized to either a combined therapist guided Internet-CBT for insomnia and depression, or to Internet-CBT for depression with an addition of a placebo intervention for insomnia. The primary purpose is to evaluate changes in insomnia and depression severity for the combination treatment compared to the depression treatment, after treatment and at 6 and 36 months follow up. A secondary purpose is to evaluate cognitive functioning before and after treatment, as well as cost effectiveness. Recruitment is done in the Stockholm County through mass media and the Internet psychiatry clinic's regular patient recruitment.

Trial 2 includes patients with insomnia who do not meet criteria for major or minor depression. All participants start therapist guided Internet-CBT for insomnia. After 4 weeks patients that are judged to be at risk of treatment failure are randomized to either continued treatment or treatment with added support intended to enhance outcome. The primary purpose is to evaluate change in insomnia severity for participants who get added support, compared to continued treatment with regular support level. A secondary purpose is to evaluate cognitive functioning before and after treatment, as well as cost effectiveness. Recruitment is done in the Stockholm County through mass media and the Internet psychiatry clinic's regular patient recruitment.

NOTE:

The first participants in trial 1 will be regarded as pilots, due to problems with the experimental treatment: technical issues as well as problems with the design of treatment modules. These problems were corrected when discovered. 12 participants in the experimental arm were affected by these errors. The pilot participants will not be included in the main analyses of data. This was decided upon on 31st of October 2014.

ELIGIBILITY:
Inclusion Criteria:

* Clinical level of Insomnia (more than 10 on ISI)
* Meets criteria for Insomnia according to DSM-IV-TR
* Enough language skills
* Only Trial 1: Meets criteria for Major or Minor Depressive Disorder according to DSM-IV-TR (for minor depression a MADRS-S-level of >19 is required).

Exclusion Criteria:

* Sleep disorders requiring other treatment
* Alcohol/drugs abuse
* Started to use or changed the dose of antidepressant drug during the last 2 months
* Somatic or psychiatric conditions requiring acute care
* Working night shifts
* Only Trial 2: Meets criteria for Major or Minor Depressive Disorder according to DSM-IV-TR (for minor depression a MADRS-S-level of >19 is required for exclusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Change (from baseline) in Insomnia Severity Index (ISI) | 0, 6 and 36 months after treatment
  7-item, self-rated questionnaire measuring change in insomnia severity. Bastien, C. H., Vallières, A., & Morin, C. M. (2001). Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Medicine, 2, 297-307.
Change (from baseline) in Montgomery Asberg Depression Rating Scale, MADRS-S | 0, 6 and 36 months after treatment
  Defined as secondary outcome measure in Trial 2. The use of two primary outcomes in trial 1 is motivated since participants have both diagnoses and the purpose is to look at effects on both insomnia and depression.
  The MADRS-S is a 9-item self-rated measure of change in depression severity. It also screens for suicidality.
  Mattila-Evenden, M., Svanborg, P., Gustavsson, P., & Åsberg, M. (1996). Determinants of self-rating and expert rating concordance in psychiatric out-patients, using the affective subscales of CPRS. Acta Psychiatr Scand, 94, 386-396.

SECONDARY OUTCOMES:
Change (from baseline) in Sleep Diary | Directly after treatment
  One week of self-ratings on a number of sleep parameters, resulting in measures of sleep latency, total sleep time, sleep efficacy, number of nighttime awakenings, subjective sleep quality and daytime functioning.
Changes (from baseline) in Actigraph data | Directly post treatment
  An actigraph is placed on the participant's arm for one week. They measure participants' activity in the form of movements. It will be used for acquiring sleep data and calculate sleep latency, total sleep time, sleep efficacy, number of nighttime awakenings and daytime activity.
Change (from baseline) in Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P) | 0, 6 and 36 months after treatment
  Health economic questionnaire evaluation cost for health care, absence of work capacity and related costs.
  Hakkaart-Van Roijen, L.,Van Straten, A., & Donker, M. (2002). Manual: Trimbos/iMTA Questionnaire for Costs Associated with Psychiatric Illness. Rotterdam: Erasmus University
Change (from baseline) in Cognitive functioning | Directly at post-treatment
  Computer based testing of executive functions, concentration, speed and memory.
Change (from baseline) in EuroQuol. EQ-5D | 0, 6 and 36 months after treatment
  General quality of life measure to complement the TIC-P in health economic analysis.
  Hinz, A., Klaiberg, A., Brahler, E., & Konig, H.H. (2006). The Quality of Life Questionnaire EQ-5D: modelling and norm values for the general population. Psychother.Psychosom.Med.Psychol., 56, 42-48.
Change (from baseline) in Sheehan Disability Scale | 0, 6 and 36 months after treatment
  Measures daily life functioning. Sheehan, D. V. (1983). The Anxiety disease. Scribner: New York
Change (from baseline) in Clinical Outcome in Routine Evaluation - 10, CORE-OM | 0, 6 and 36 months after treatment
  Measures psychological health in general. Evans, C., Connell, J., Barkham, M., Margison, F., McGrath, G., Mellor-Clark, J. & Audin, K. (2002). Towards a standardised brief outcome measure: psychometric properties and utility of the CORE-OM. The British journal of psychiatry : the journal of mental science 180, 51-60.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Kaldo, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Internetpsykiatrienheten (Internet Psychiatry Clinic) Psykiatri Sydväst, SLSO, Stockholm, Sweden

REFERENCES:
- [Derived] Tamm S, Jernelov S, Forsell E, Eldh A, Hallek de Oliveira A, Maurex L, Kaldo V, Blom K. Objectively measured cognitive function in insomnia patients with and without comorbid depression treated with cognitive behavioral therapy for insomnia. BMC Psychiatry. 2025 Oct 2;25(1):916. doi: 10.1186/s12888-025-07460-5. PMID 41039374
- [Derived] Kraepelien M, Blom K, Forsell E, Hentati Isacsson N, Bjurner P, Morin CM, Jernelov S, Kaldo V. A very brief self-report scale for measuring insomnia severity using two items from the Insomnia Severity Index - development and validation in a clinical population. Sleep Med. 2021 May;81:365-374. doi: 10.1016/j.sleep.2021.03.003. Epub 2021 Mar 16. PMID 33813233
- [Derived] Forsell E, Jernelov S, Blom K, Kraepelien M, Svanborg C, Andersson G, Lindefors N, Kaldo V. Proof of Concept for an Adaptive Treatment Strategy to Prevent Failures in Internet-Delivered CBT: A Single-Blind Randomized Clinical Trial With Insomnia Patients. Am J Psychiatry. 2019 Apr 1;176(4):315-323. doi: 10.1176/appi.ajp.2018.18060699. Epub 2019 Jan 30. PMID 30696270
- See also: The public page of the Internet Psychiatry Clinic — http://www.internetpsykiatri.se